CLINICAL TRIAL: NCT03872830
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-exploratory Phase II Clinical Trial to Evaluating the Efficacy and Safety of Felbinac Trometamol Injection in the Treatment of Moderate to Severe Pain After Surgery
Brief Title: A Phase Ⅱ Clinical Study Trial of Felbinac Trometamol Injection in China
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BALF-PAIN-2001
Record Dates: First submitted 2019-03-06; First posted 2019-03-13 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: group1 (Experimental): Generic name:Felbinac Trometamol Injection; Placebo:normal saline Dosage form:Injection Dosage:47.13mg Volume:2ml Frequency:Multi-dose Duration:1 day. A total of 40 subjects,40 received the test drug .
  Interventions: Drug: Felbinac Trometamol Injection
- Experimental: group2 (Experimental): Generic name:Felbinac Trometamol Injection; Placebo:normal saline Dosage form:Injection Dosage:94.25mg Volume:4ml Frequency:Multi-dose Duration:1 day. A total of 40 subjects,40 received the test drug .
  Interventions: Drug: Felbinac Trometamol Injection
- Experimental: group3 (Experimental): Generic name:Felbinac Trometamol Injection; Placebo:normal saline Dosage form:Injection Dosage:188.5mg Volume:8ml Frequency:Multi-dose Duration:1 day. A total of 40 subjects,40 received the test drug .
  Interventions: Drug: Felbinac Trometamol Injection
- Experimental: group4 (Placebo Comparator): Generic name:Placebo; Placebo:normal saline Dosage form:Injection Dosage:4ml/injection Volume:10ml Frequency:Multi-dose Duration:1 day. A total of 40 subjects,40 received the placebo.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Felbinac Trometamol Injection — Felbinac Trometamol Injection diluted to 100 ml with 0.9% sodium chloride injection,a 30-minute period using a Microinjection pump.
  One dose at 8h and 16h after the start of the first dose,the first intravenous infusion was started at the end of the operation (Skin suture completes the last stitch).the drug was given 3 times,3 times/day,once every 8 hours.
  Arms: Experimental: group1; Experimental: group2; Experimental: group3
Drug: Placebos — Placebo diluted to 100 ml with 0.9% sodium chloride injection,a 30-minute period using a Microinjection pump.
  One dose at 8h and 16h after the start of the first dose,the first intravenous infusion was started at the end of the operation (Skin suture completes the last stitch).the drug was given 3 times,3 times/day,once every 8 hours.
  Arms: Experimental: group4

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, dose-exploratory phase II clinical trial to evaluating the efficacy and safety of Felbinac Trometamol Injection in the treatment of moderate to severe pain after surgery.Main purpose is preliminary evaluation the effectiveness of Felbinac Trometamol Injection in the treatment of moderate and severe pain after surgery.Secondary purpose is to explore the dosage regimen of Felbinac Trometamol Injection in the treatment of moderate and severe pain after surgery, and provide data support for later clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 18≤age≤65 years of age, gender is not limited;
* ASA grade I or II;
* 18 ≤ body mass index (BMI) ≤ 30 [BMI = weight (kg) / height 2 (m2)];
* Inpatients who underwent open surgery under elective general anesthesia (including gallbladder, intestinal or lower abdominal surgery, etc.), or laparoscopic surgery with a single surgical incision ≥ 5 cm;
* Expected to require more than 24 hours of PCIA( patient controlled intravenous analgesia) treatment after surgery ;
* Ability to understand research procedures and pain scales, operate PCIA devices, and communicate effectively with researchers;
* Agree to participate in the trial and voluntarily sign the informed consent form.

Exclusion Criteria:

* Those who have a history of chronic pain for more than 3 months or who are undergoing regular analgesia for more than 3 months;
* Those who used other analgesics, muscle relaxants or sedatives within 24 hours before operation (excluding those required for this operation), or those who used long-acting non-steroidal anti-inflammatory drugs (NSAIDs) within 12 hours, or those who used short-acting non-steroidal anti-inflammatory drugs (NSAIDs) within 6 hours before operation(See Annex 1).
* A person with high bleeding risk, and also including who with congenital bleeding disorders (such as hemophilia), thrombocytopenia (PLT < 80 × 10 ∧ 9 / L), abnormal platelet function (such as idiopathic thrombocytopenic purpura, disseminated intravascular coagulation, congenital platelet dysfunction, etc.) or any clinically significant active bleeding, coagulopathy;
* A person who received full-dose anticoagulant therapy, activated protein C or thrombolytic drugs within 6 hours before surgery (except for heparin subcutaneous injection for preventive treatment);
* People with heart failure (NYHA grade III or IV), unstable angina pectoris, acute myocardial infarction, and severe arrhythmia within 6 months before surgery
* Hypertensive patients who have not been satisfactorily controlled by blood pressure (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥105mmHg), or ACEI/diuretics for ≥30 days, or hypotension (systolic blood pressure <90mmHg);
* People with bronchial asthma, pulmonary heart disease or other serious respiratory diseases;
* Person with gastrointestinal ulcer and a history of gastrointestinal bleeding 6 weeks before operation and required medical treatment;
* Those with previous cerebral arteriovenous malformations, cerebral aneurysms, brain tumors, or preoperative traumatic brain injury, intracranial surgery, history of stroke;
* Patients with poor glycemic control of diabetes (random blood glucose > 11.1mmol / L);
* Patients with autoimmune diseases, connective tissue diseases, etc. who need long-term use of adrenocortical hormone therapy;
* Abnormal liver and kidney function: ALT/AST> 2 times the upper limit of normal value, or creatinine> upper limit of normal value, or dialysis treatment within 28 days before surgery;
* Allergic constitution, or known to be allergic to this drug, NSAIDs, and opioids;
* Patients who are afflicted with narcotic drugs, drugs, or resistant to opioids;
* A woman who is breast-feeding or pregnant, who is unable or unwilling to follow the investigator's guidance during the study period and within 3 months after the last study treatment;
* Those who have participated in other clinical trials within 3 months before surgery;
* Investigators believe that it is not suitable for participating in this research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
24h total morphine consumption | up to 24hours after multi-dose
  The the total amount of morphine within 24 hours after the end of first drug administration

SECONDARY OUTCOMES:
Area under the pain intensity curve(AUC) | up to 24 hours after multi-dose
  Pain intensity under exercise/rest state - area under the time curve
Press time | up to 24 hours after multi-dose
  The first time to press the analgesic pump for analgesia
Total number of analgesia pump presses | up to 24 hours after multi-dose
  Total number of analgesic pump presses within 24 hours after the first dose
The number of effective presses of analgesia pump | up to 24 hours after multi-dose
  The number of effective presses of analgesia pump within 24 hours after the end of the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Wen Ouyang, MD, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- Shijiazhuang Yiling Pharmaceutical Co.,Ltd, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No